CLINICAL TRIAL: NCT04837534
Title: Effect of Counseling and Reminders in Improving the Follow-up Rate of Pediatric Patients (0-16 Years) at Bharatpur Eye Hospital, Nepal: an Intervention Study
Brief Title: Improving the Follow up Rate for Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seva Foundation (Other)
Collaborators: Bharatpur Eye Hospital (Other); Indian Institute of Public Health, India (Other); Seva Canada Society (Other); Queen's University, Belfast (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BEH/ERB/761/2020 P
Record Dates: First submitted 2021-03-31; First posted 2021-04-08 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: CNLDO - Congenital Nasolacrimal Duct Obstruction; Amblyopia; Conjunctivitis; Eye Injuries; Corneal Ulcer; Strabismus
Keywords: Follow up; Counselling; SMS and phone calls; intervention study; Children; Peadiatric eye conditions
MeSH Terms: conditions — Amblyopia; Conjunctivitis; Eye Injuries; Corneal Ulcer; Strabismus | interventions — Spermine Synthase

STUDY DESIGN:
Intervention Model Description: Primary Purpose: Our primary objectives are a) to determine if parental counseling has an impact on adherence to follow-up, b) To determine if reminders through phone calls and SMS increase the follow-up rate in pediatric patients.
  Assessing the cost-effectiveness of counseling and reminder SMS and phone calls, and determining the role of counselors and their sustainability are our secondary objectives. We hypothesize that counseling will increase the follow-up rate from 22% to 50% and reminders through phone calls and SMS from 22% to 25% of pediatric patients attending Bharatpur Eye Hospital
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Counseling group (Experimental): In this group after the children have been examined, treatment plan and follow up schedule been advised by a pediatric ophthalmologist, parents/guardians along with the child will receive counseling from a trained counselor as per the set counseling protocol in every follow-up visits and will also be provided with the disease-specific information leaflets as an additional information material before the child is discharged from the department.
  Interventions: Behavioral: Counseling group
- SMS and phone call reminder group: (Experimental): In this group after the children have been examined, treatment plan and the follow-up schedule been advised, they will be discharged from the department but later they will receive reminders through short messaging text (SMS) and phone calls as per the set protocol
  Interventions: Behavioral: SMS and phone call reminder group
- Routine standard care group (No Intervention): In this group, the children will undergo ocular examination, and treatment plan. They will be discharged from the department and advised accordingly including a routine follow-up schedule as per hospital protocol.

INTERVENTIONS:
Behavioral: Counseling group — In this group after the children have been examined, treatment plan and follow up schedule been advised by a pediatric ophthalmologist, parents/guardians along with the child will receive counseling from a trained counselor as per the set counseling protocol in every follow-up visits and will also be provided with the disease-specific information leaflets as an additional information material before the child is discharged from the department.
  Arms: Counseling group
Behavioral: SMS and phone call reminder group — In this group after the children have been examined, treatment plan, and the follow-up schedule been advised, they will be discharged from the department but later they will receive reminders through short messaging text (SMS) and phone calls as per the set protocol.
  Arms: SMS and phone call reminder group:

SUMMARY:
Follow-up of pediatric patients is important for their regular ocular morbidity monitoring, especially for amblyopia management. An observatory data of 1st week (1st to 7th) of January 2019 revealed that the follow-up compliance was very low (22%) among children aged 0-16 years in the pediatric department of Bharatpur Eye Hospital. A problem tree analysis showed a lack of awareness in children and their parents regarding the importance of follow-up and patients forgetting regarding the follow-up visit, usually when there is the long duration of follow up are the major contributing factors for poor adherence to follow-up. So, an intervention study was aimed at finding the effectiveness of counseling and reminders through SMS and phone calls to improve the follow-ups.

All pediatric patients 0-16 years of age with ocular conditions requiring at least 3 follow-ups in the study period (January 2021 to April 2021) will be included. Two hundred and sixty-four participants will be equally distributed to three groups: routine standard care, counseling, and reminders with SMS and phone calls. In the routine care group, children will undergo routine care as per existing practice in the hospital and there will be no additional intervention. In counseling group, in addition to routine care parents/guardians along with the child will receive counseling from a trained counselor as per the set counseling protocol in every follow-up visits and will also be provided with the disease-specific information leaflets as additional information material before the child is discharged from the department. In the SMS and phone call reminder group, in addition to routine care, parents/guardians of children will receive reminders through short messaging text (SMS) 3 days and phone calls one day prior to the scheduled visit.

Compliance to follow up Participants completing all the three follow-up visits as per the schedule within the window period of +/-2 days will be considered as a complaint to follow up. However, the follow-ups of all the participants will be recorded although that is beyond the window period. The primary outcome will be measured by the proportion of children completing all three scheduled follow-ups.

The ethical approval has been obtained from the Institutional Review Committee of NHRC (ERB protocol registration number 761/2020 P). Informed consent will be taken from parent and child.

Conclusion:

If interventions improve the follow-up rate and are cost-effective, this can be applied in all the departments of the hospital.

DETAILED DESCRIPTION:
Need: Childhood visual impairment and blindness remains an important public health issue. It is estimated that around 14 million children in the world are blind. Nepal Pediatric Ocular Disease study found that prevalence of blindness and visual impairment in the community was 0.068% (95% CI 0.02%-0.12%) and 0.097% (95% CI 0.04%-0.15%) respectively. Increasing the global knowledge base for planning for childhood eye care services is a top priority in order for children with visual impairment to realize their full visual potential. Follow-up of pediatric patients is important for their regular ocular morbidity monitoring, especially for amblyopia management. A study done in India revealed distance and cost as major barriers, as was the inability of the eye care center to communicate the importance of follow-up. Another study done in Nepal found poor follow-up rates for post-cataract surgery patients which however improved after implementation of a post-operative follow-up program.

Bharatpur Eye Hospital observed that there is poor adherence to follow-up visits. An observatory data of 1st week (1st to 7th) of January 2019 revealed that the follow-up compliance was very low among children aged 0-16 years in the pediatric department. Among the children advised for follow up only 22% were found to have come for at least one follow-up visit. Therefore, there was the need to implement measures to improve the follow-up rate.

Potential impact: High-quality pediatric counseling service, follow-up program, tracking system, and cell phone reminders resulted in the improved follow-up of pediatric patients in Lumbini Eye Institute, Nepal.6 Many studies have compared different methods of reminder options like telephone calls, email, SMS in order to improve the compliance to followup.7,8,9,10. Bharatpur Eye Hospital aims to find the effectiveness of counseling and reminders through SMS and phone calls on improving the follow-up rates of pediatric patients.

Bharatpur Eye Hospital assumes that with the proposed intervention the follow-up rate would increase to 50% considering the similar increase in follow-up rate in postoperative cataract surgery patients done in Lumbini Eye Institute (around 20% increase in follow up)6. In addition to it, another study done in London showed the use of SMS reminders for ophthalmology outpatient appointments reduced the non-attendance rates by 6.9%.18Improving follow-ups of patients is important to meet the treatment goal and provide effective and complete treatment for particular ocular problems. Adherence to follow-up is even more vital for children because the visual system is still in the developing phase in young children and loss of follow-up may lead to loss of vision. So, for quality treatment, patient satisfaction and improvement of the visual status of children, and revenue generation for the hospital it should be the priority area for the hospital to find ways for improving the existing low adherence to follow up in pediatric patients.

Study site: Bharatpur, Chitwan is located in the central part of the country, which is 150 K M. west from Kathmandu and 130 K. M. east from Lumbini (Bhairahawa) with an area of 2218 sq. Kilometer. The hospital, named Bharatpur Eye Hospital is located in the delightful city of Bharatpur, the capital of Chitwan district, by the bank of Narayani River, a place of pilgrimage of the Hindus. It is a tertiary eye hospital that ranks first among the eye hospitals in Nepal.

Study population: All pediatric patients 0-16 years of age attending the pediatric department of Bharatpur Eye Hospital from January 2021 to April 2021. In the pediatric department children aged 0-16 years are being examined as per the hospital policy although younger than 18 years is considered as children as per WHO.

Eligibility: Enrolment criteria: all pediatric patients 0-16 years age attending Bharatpur Eye Hospital and advised for at least 3 follow up visits within 4 months period (January 2021 to April 2021)

Sample size: A sample size of 264 (88 in each of the three groups) pediatric patients will be targeted with an adjusted significance level of 0.02, 80% power, and 10% loss to follow up. The sample size for comparison of two proportions using Bonferroni correction (level of significance=0.05/k=3 comparisons) was adopted. The proportion of attendance in counseling (p1) and reminder SMS/phone call(p2) are taken as 50% (0.5) and 25% (0.25) respectively.

The sample size has been calculated as per the general objective that "To determine the effect of counseling and reminders through SMS and phone calls in improving the follow-up rates in pediatric patients". Hence this study is not exclusively looking at the difference between counseling and reminder through SMS and phone call with routine standard care group separately. That means the project is looking for overall improvement in follow-up rate based on the package of the interventions vs routing standard care group. For ease of understanding 2 groups have been created among the intervention group.

Randomization: None Program: The total costs involved in implementing the interventions will be compared with the attendance of follow-up patients and the revenue generated through their follow-ups. The intervention costs include the salary for the team members. In addition to the costs for the phone calls and reminder SMS telecommunication charges, the cost for equipment, stationary, and the charges for utility services like water and electricity will also be included as the cost for implementing interventions. Cost-effectiveness will be analyzed separately for counseling and reminders (phone &SMS) by calculating the total cost incurred per attendance of follow-up in each intervention group and the total revenue generated through the attendance.

Data collection: Records of the participants from the first visit to all the follow-up visits will be maintained in the department by the Assistant of Pediatric Ophthalmologist. In order to obtain the required data from the participants, a proforma has been designed based on variables pertaining to sociodemographic and follow-up. Proforma has been developed in the English language, sequence of questions will be carefully looked into as well as skips pattern (if any). Questions pertaining to identification and socio-demographic information appeared first, then follow-up points.

The record of the patients will be kept even if they come for follow-up beyond the set window period (+/- 2 days), however in this case they will not be considered compliant to follow up.

The assistant will also assign the group to the patients (if they receive any intervention or not) as per the study procedure.

Data management plan: A follow-up recording file (3 in number, one each for routine standard care, counseling, and reminders through SMS and phone call) will be maintained. These follow-up details will also be entered in the excel sheet on the same day as a backup in case the paper records are lost or destroyed. The entry of all the details from the proforma will be done in the excel sheet by the assistant and the status of record maintenance will be regularly monitored. The data entry program will be designed in the SPSS version (The latest version). Mr. Gopal, who is an optometrist and Co-PI in this study, will do the first and second data entries. Validation of the two data sets will be done. Corrections will be made where required by comparing the computer data file with the original proforma.

The local statistician will also be part of this study

Data analysis plan: Data will be processed and analyzed using SPSS latest version

Descriptive analysis:

In the first step descriptive analysis will be done, summarizing demographic variables by computing means with standard deviation for continuous variables and percentages for categorical variables. Amputation and intention to treat analysis will also be conducted (if required).

Univariate analysis:

Univariate logistic regression analysis will be conducted by comparing two variables for each variable of interest using odds ratio (OR) and their 95% confidence intervals (CI). Likelihood ratio test will be used to estimate odds ratio and 95% CI for odds ratio for all associations of interest.

Multivariate analysis:

Multivariate logistic regression analysis will be performed to adjust for simultaneous effects of multiple factors on the outcome variable. The criteria for inclusion of factors in the multivariate analysis are to include all variables from the univariate analysis with a p-value of <= 0.1 along with all the variables of known biological importance. To assess the importance of each variable included in the model, a Wald statistic for each variable will be used.

Before conducting multivariate analysis, the association among independent variables will be checked by the chi-square test. For independent variables having more than two categories, dummy variables will be created. All the variables meeting the above selection criteria will be entered one by one, starting with the highly significant factor from the univariate analysis. The overall significance of independent variables in the model will be assessed by the likelihood ratio test (G statistic). The selection of the final model will be based on parsimony, biological interpretability, and statistical significance. The parameters of the logistic regression model will be estimated by the maximum likelihood method. The adjusted odds ratios (ORs) and their 95% confidence intervals (CIs) will be computed using the estimates of parameters of the final model. The dependent variable will be dichotomous, either follow-up rate increased or as it is (no difference). The final model will be tested for goodness-of-fit by Hosmer- Lemeshow chi-square (x2) statistic. P-values will be noted to assess the model fit.

Monitoring: Supervision and monitoring will be done by PI and co-PI every week to check the study participants' enrolment, record keeping, and maintenance of data and ensure research activities are taking place as per the research protocol.

Ethics and consent: The ethical approval for the study will be obtained from the Review Committee of NNJS / Nepal Health Research Council. Written consent will be taken from the children in an assent form (if 9 years or older) and from their parents/guardians in a consent form before enrolling them in the study. Approval for conducting the study has also been taken from Bharatpur Eye Hospital.

ELIGIBILITY:
Inclusion Criteria:

* all pediatric patients 0-16 years age advised for at least 3 follow up visits within 4 months period (January 2021 to April 2021) at Bharatpur Eye Hospital
* Patients who require weekly, bi-weekly (fortnight), or monthly follow up visits,
* In certain conditions, some severe cases require earlier follow up than the scheduled follow up schedule, those cases will be included,
* Parents/guardians of children who own a mobile phone or have daily access to a phone and are able to use the SMS (Short Message Sending) feature on these phones,
* Parents of children willing to enroll their children in the study

Exclusion Criteria:

* Children who require less than 3 follow up visits,
* Ocular conditions requiring daily follow up visits will be excluded because it is not feasible to send the reminder phone call and SMS for daily follow up
* Children who have already been treated and under regular follow up,
* Children with ocular conditions requiring to follow up beyond four months,
* Children whose follow up schedules fall beyond the study duration,
* Parents/ guardians of the children not willing to participate in the study.

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 264 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Proportion of children completing all three follow up visits | 4 months
  The primary outcome is the proportion of children completing all three follow up visits in routine standard care group, counseling group and reminders through SMS and phone call group.

SECONDARY OUTCOMES:
Factors affecting compliance to follow-up | 2 months
  1. effect of parental/guardian education status in compliance to follow-up,
  2. visual status of the children in subsequent follow-up visit, c)effect of travelling distance and cost in compliance to follow-up.
Cost-effectiveness of the intervention | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Dr Manisha Shrestha, Principal Investigator — Bharathpur Eye Hospital
Locations (1):
- Bharatpur Eye Hospital, Bharatpur, Chitwan, Nepal

REFERENCES:
- [Derived] Shrestha M, Bhandari G, Kamalakannan S, Murthy GVS, Rathi SK, Gudlavalleti AG, Agiwal V, Pant H, Pandey B, Ghimire R, Ale D, Kayastha S, Karki R, Chaudhary DS, Byanju R; Operational Research Capacity Building Study Group. Evaluating the Effectiveness of Interventions to Improve the Follow-up Rate for Children With Visual Disabilities in an Eye Hospital in Nepal: Nonrandomized Study. JMIR Pediatr Parent. 2023 Feb 23;6:e43814. doi: 10.2196/43814. PMID 36821366
- [Derived] Shrestha M, Bhandari G, Rathi SK, Gudlavalleti AG, Pandey B, Ghimire R, Ale D, Kayastha S, Chaudhary DS, Byanju R; Operational Research Capacity Building Study Group. Improving the Follow-up Rate for Pediatric Patients (0-16 years) of an Eye Hospital in Nepal: Protocol for a Public Health Intervention Study. JMIR Res Protoc. 2021 Oct 8;10(10):e31578. doi: 10.2196/31578. PMID 34521615